CLINICAL TRIAL: NCT04356820
Title: The Effect of Music Played and Acupressure Application on Pain and Anxiety in Women Undergoing Gynecological Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Didem Kucukkelepce, Didem Kucukkelepce, Adiyaman University Research Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Adıyaman_Universty
Record Dates: First submitted 2020-04-16; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Pain, Acute; Anxiety Acute
Keywords: acupressure,; nursing; music; gynecological examination
MeSH Terms: conditions — Acute Pain | interventions — Acupressure; Music Therapy

STUDY DESIGN:
Intervention Model Description: randomized
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acupressure (Experimental)
  Interventions: Other: acupressure
- music (Experimental)
  Interventions: Other: acupressure
- control (No Intervention)

INTERVENTIONS:
Other: acupressure — Data collection took about 10 to 15 minutes. Then the woman invited to the examination room was asked to pull one of the envelopes with the names of the groups. The women who pulled the acupressure envelope were given a semi-sitting position where the acupressure application can feel comfortable and the researcher can easily apply the acupressure points. Before the acupressure application, massage was applied for 30 seconds to ensure circulation. Afterwards, 90 seconds consecutive pressures were applied to the specified acupressure points in a certain order (SP 6, Li 4), taking into account the direction of the meridian. After the examination, the pain formed during the gynecological examination was evaluated by applying the Short Form-McGill Pain Questionnaire without leaving the examination room
  Other Names: music
  Arms: acupressure; music

SUMMARY:
This study was carried out to determine the effect of listening to music and acupressure application in reducing pain and anxiety during gynecological examination.

ELIGIBILITY:
Inclusion Criteria:

* - not to be pregnant,
* no hearing problems
* Being between the ages of 19 and 65, Not having any psychiatric illness,
* No gynecological cancer, Not to have any deformity in her extremities

Exclusion Criteria:

-

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 156 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
questionnaire and scale | 12 weeks
  McGill pain scale was developed by Melzack in 1987 and its validity and reliability in Turkish Yakut et al. (2007). In this study, the Short Form-McGill Pain Questionnaire (KF-MAA), whose validity and reliability was used and frequently used by Biçici (2010), was applied. This questionnaire consists of a total of 15 descriptive words to determine the sensory (11 words) and affective (4 words) dimensions of pain. In this section, the severity of pain (0 = none, 1 = mild, 2 = moderate, 3 = severe) is evaluated and three pain scores (sensory, affective and total pain rate = sensory affective) are obtained. In addition, the pain felt at the time of measurement is measured with the Visuel Analog Scale (VAS) and the total pain intensity is measured with a 6-point Likert scale. On this scale, 0 = no pain, 1 = mild, 2 = disturbing, 3 = distressing, 4 = terrible, 5 = unbearable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Didem Simsek Kucukkelepce, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No